CLINICAL TRIAL: NCT06775457
Title: Genome Analysis of Human Endogenous Retroviruses (HERVs) and Gut Microbiota in Patients With SARS-CoV-2 Infection, Kawasaki Disease and Other Febrile and Inflammatory Diseases With Systemic Involvement in Pediatric Age.
Brief Title: Genome Analysis of Human Endogenous Retroviruses (HERVs)(COVID19)
Acronym: HERV_COVID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HERV_COVID
Record Dates: First submitted 2024-12-01; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: SARS CoV-2; Kawasaki Disease; Retrovirus Infection
Keywords: SARS-COV2; Kawasaki Disease; Human Endogenous Retroviruses
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Retroviridae Infections | interventions — Specimen Handling

STUDY DESIGN:
Intervention Model Description: In vitro prospective, nongenetic human tissue study on biological specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): The study will be offered consecutively to each patient in whom Kawasaki Disease, Schonlein-Henoch purpura, symptomatic SARS-CoV-2 infection, febrile virosis, and with inflammatory diseases with systemic involvement are diagnosed.
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — Blood samples and fecal samples will be taken from patients during evaluation visits. Blood samples will be analyzed for the study of HERVs. While fecal samples will be analyzed for the characterization of gut microbiota.

SUMMARY:
Human Endogenous Retroviruses (HERVs) are ancient sequences that became integrated into our DNA during evolutionary processes.

The significance of their presence in DNA is still being studied, but HERVs appear to be involved in the regulation of the immune response.

The gut microbiota is the set of microorganisms that physiologically colonize the gastrointestinal tract. Progressively increasing attention is being paid to the gut microbiota and its potential role in diseases of various kinds. In particular, it has recently been shown how abnormalities in the microbiota can affect immune regulation by determining the occurrence of certain diseases. One objective of the study is to evaluate whether there is an association between the expression of HERVs and clinical manifestations in pediatric age in patients with various diseases such as Kawasaki Disease, IgA Vasculitis/Schonlein-Henoch's Purpura, SARS-CoV-2 infection, or, finally, febrile virosis.

Another objective of the study is to evaluate whether there is an association between the presence of particular types of bacteria in the gut microbiota and clinical manifestations in pediatric age in patients with Kawasaki Disease, IgA Vasculitis/Schonlein-Henoch purpura, SARS-CoV-2 infection or febrile virosis.

The results from this may open new perspectives for both the care and therapeutic management of children with these diseases.

DETAILED DESCRIPTION:
The literature provides us with indications that HERVs have been found to be implicated in the pathogenesis of numerous complex diseases, characterized by a multifactorial etiology on a genetic susceptibility basis. Indeed, it is hypothesized that HERVs may represent the link between genetic risk factors and infectious/environmental factors, thus contributing to the onset and/or progression of these diseases. It has also been pointed out that there is an interaction between HERVs and cytokines, in that reactivation of HERVs appears to shape the innate immune response, evoking the production of pro-inflammatory cytokines, and conversely, inflammatory effectors could in turn be responsible for further increasing HERVs activity. A similar point can be made regarding the gut microbiota and its potential role in modulating both innate and adaptive immune responses.

An imbalance of gut microbiota (GM), thus of host-GM homeostasis, as a result of various environmental stimuli ( antibiotic intake, diet, geographic area...), may alter the immune system response favoring in some cases an aberrant immune response by modulating the innate and adaptive immune system (IS). It can influence inflammasome function in innate immune cells and enterocytes, either through a direct interaction between GM and immune cells, or through the production of metabolites (lipopolysaccharides, peptidoglycans, microbial nucleic acids, glucans, and mannans) that regulate IS function. Short-chain fatty acids, produced by fermentation of lipopolysaccharides from GM exert an important role on the host IS: butyrate modifies the cytokine production profile of helper T cells and promotes the integrity of the intestinal epithelium, while acetate promotes the resolution of intestinal inflammation. Based on this rationale, we intend to conduct a study of patients with Kawasaki disease (KD), IgA vasculitis/Schonlein-Henoch purpura, SARS-CoV-2 infection, and febrile virosis in pediatric age. Particularly in Kawasaki disease, the study could identify in HERVs a causative/favorable role in disease onset and identify individuals at higher risk of severe form in terms of cardiac injury and response to conventional therapy, and contribute the identification of possible new therapeutic targets. The increased expression of HERVs could, in fact, identify subjects at higher risk for a severe form, who could benefit from additional personalized therapy early on and closer cardiologic instrumental follow-up for coronary lesions. Relative to IgA vasculitis/Schonlein-Henoch purpura, determination of altered transcriptional activity of HERVs in affected subjects could help define a prognostic factor of severe pictures. We also intend to compare the characteristics of affected subjects with those of KD patients, given the vasculitic nature of both diseases, to highlight differences or similarities in expression. In pediatric SARS-CoV-2 infection, we believe that the study of the expression of HERVs may be a useful aid in explaining the increased susceptibility of some individuals to development of severe disease pictures, especially the development of MIS-C picture. In inclusion of subjects with significant febrile virosis pictures, such as to require hospitalization, is aimed both at identifying possible patterns of predisposition for the development of systemic pictures in the context of viral infections and to compare clinical-laboratory features with respect to patients with symptomatic SARS-CoV-2 infection. Similarly, in each of the categories of patients previously described, we believe that analysis of GM can help determine whether particular profiles and characteristics may condition different disease pictures through modulation of immune response and by maintaining intestinal mucosal integrity.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, newly diagnosed with Kawasaki disease
* Pediatric patients, newly diagnosed with Vasculitis
* Pediatric patients, newly diagnosed with SARS-CoV-2 infection
* Pediatric patients, newly diagnosed with febrile virosis
* Pediatric patients with inflammatory diseases with systemic involvement

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HERVs analysis | through study completion, an average of 1 year
  Investigate the expression levels of specific HERVs families in PBMCs of patients with Kawasaki disease, IgA vasculitis/Schonlein-Henoch purpura, SARS- CoV-2 infection, and febrile virosis and inflammatory diseases with systemic involvement in pediatric age.
Microbiota characterization | through study completion, an average of 1 year
  Characterize the MI composition of subjects with Kawasaki disease, IgA vasculitis/Schonlein-Henoch's purpura, SARS-CoV-2 infection, and febrile virosis and inflammatory diseases with systemic involvement in pediatric age included by culture-independent method (16S rRNA gene sequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Fabi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (5):
- Italy (5):
  - Ospedale Ramazzini di Carpi, Azienda USL di Modena UO Pediatria, Carpi, Modena
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve ed Intensiva, Bologna
  - Azienda Ospedaliera-Universitaria di Modena, Modena
  - IRCCS Ospedale Pediatrico Bambino Gesù UOC Pediatria Generale, Roma
  - Ospedale Regina Margherita, Torino, UO Reumatologia Pediatrica, Torino